CLINICAL TRIAL: NCT06432088
Title: Prospective, Multi-center, Single-arm, Open Label Study Designed to Assess the Safety and Feasibility of Liver Retraction With the Levita Magnetic Surgical System: Extended Magnetic Grasper Device
Brief Title: Safety and Feasibility of Liver Retraction With the Levita Magnetic Surgical System: Extended Magnetic Grasper Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LVT009; CP009 (Other: Levita Magnetics)
Record Dates: First submitted 2024-05-16; First posted 2024-05-29 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery Candidate; Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extended Magnetic Grasper Device (Experimental): Evaluation of the safety and effectiveness of the Extended Magnetic Grasper Device in patients undergoing bariatric and/or hiatal hernia procedures, as a liver retractor grasping the liver and/or the tissue surrounding the crus of the diaphragm.
  Interventions: Device: Extended Magnetic Grasper Device

INTERVENTIONS:
Device: Extended Magnetic Grasper Device — The purpose of this study is to evaluate the safety and effectiveness of the Extended Magnetic Grasper Device in patients undergoing bariatric and/or hiatal hernia procedures, as a liver retractor grasping the liver and/or the tissue surrounding the crus of the diaphragm.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Extended Magnetic Grasper Device in patients undergoing bariatric and/or hiatal hernia procedures, as a liver retractor grasping the liver and/or the tissue surrounding the crus of the diaphragm.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of the Levita Magnetic Surgical System Version 2 in patients undergoing bariatric and/or hiatal hernia procedures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Scheduled to undergo elective bariatric and/or hiatal hernia procedures.
* Willing and able to provide a written Informed Consent Form (ICF) to participate in the study prior to any study required procedures.

Exclusion Criteria:

* Individuals with pacemakers, defibrillators, or other electromedical implants.
* Individuals with ferromagnetic implants.
* American Society of Anesthesiologists (ASA) score of III or IV.
* Significant comorbidities: cardiovascular, neuromuscular, chronic obstructive pulmonary disease, and urological disease (renal failure).
* Clinical history of impaired coagulation confirmed by abnormal blood tests.
* Individuals has signs of hepatic abnormality (e.g.: cirrhosis, liver failure, increase in liver enzymes, etc.).
* Anatomical abnormality or disease of intended target tissue noted after initiation of index procedure that would prevent device use.
* Pregnant or wishes to become pregnant during the length of study participation.
* Individual is not likely to comply with the follow-up evaluation schedule.
* Participating in a clinical trial of another investigational drug or device.
* Prisoner or under incarceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santiago Oriente Dr. Luis Tisné Brousse, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Magnetic Grasper Device
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Extended Magnetic Grasper Device
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Chile | 30
BMI [Mean (Standard Deviation); unit: kg/m²] | 39.09 (5.46)

OUTCOME MEASURES:

1. Primary Outcome: Number of Device Related Adverse Events
Description: All adverse events will be captured and reported. Adverse events will be summarized by relatedness to the device and/or procedure, seriousness and level of severity.
Time Frame: 30 days
Measure: Number; unit: Device related adverse events
Arm/Group | Extended Magnetic Grasper Device
Number analyzed (Participants) | 30
Device related adverse events | 0

2. Primary Outcome: Mobilization Requiring Additional Retractors
Description: Ability to adequately mobilize the liver to achieve an effective exposure of the target tissue. Adequate mobilization is not achieved if it is necessary to use another liver retractor during the procedure.
Time Frame: 1 day
Measure: Number; unit: Procedures w/ additional retractors
Arm/Group | Extended Magnetic Grasper Device
Number analyzed (Participants) | 30
Procedures w/ additional retractors | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and serious adverse events (SAEs) were recorded from index procedure through study exit (30 day follow up).
Arm/Group | Extended Magnetic Grasper Device
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 14/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Magnetic Grasper Device (N=30)
Ecchymosis in Surgical Incision (Skin and subcutaneous tissue disorders) | 5 (5)
Liver Capsule Minor Abrasion (Surgical and medical procedures) | 5 (5)
Petechia (Skin and subcutaneous tissue disorders) | 7 (7)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Transverse Colon Injury (Gastrointestinal disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT06432088/Prot_SAP_000.pdf